CLINICAL TRIAL: NCT00853554
Title: An Open-Label, Randomized, Two-Period, Crossover Study to Evaluate the Relative Bioavailability of a Test Tablet Formulation of Hydromorphone Hydrochloride (8 mg) Compared to an Equivalent Dose of a Commercially Available Reference Drug Product (DILAUDID®, 8 mg Tablet, Knoll Pharmaceutical Company) in Normal Human Subjects Under Fasting Conditions
Brief Title: Fasting Study of Hydromorphone Hydrochloride 8 mg Tablets and Dilaudid 8 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Herbert Neuman, MD/Chief Medical Officer, Mallinckrodt
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3249-02-769
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Healthy Subjects; Bioequivalence
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Hydromorphone Hydrochloride tablet 8 mg
  Interventions: Drug: Hydromorphone Hydrochloride tablet 8 mg
- B (Active Comparator): Dilaudid® tablet 8 mg
  Interventions: Drug: Dilaudid® tablet 8 mg

INTERVENTIONS:
Drug: Hydromorphone Hydrochloride tablet 8 mg — Hydromorphone Hydrochloride tablet 8 mg, single dose fasting
  Arms: A
Drug: Dilaudid® tablet 8 mg — Dilaudid® tablet 8 mg, single dose fasting
  Arms: B

SUMMARY:
The objective of this open-label, randomized, two-period crossover study was to compare the oral bioavailability of a Mallinckrodt test tablet formulation of hydromorphone 8 mg to an equivalent oral dose of a commercially available hydromorphone tablet (DILAUDID® 8 mg, Knoll Pharmaceutical Company) in a test group of healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-lactating females, 18 years of age or older.
2. Female subjects must be postmenopausal for at least one year, or surgically sterile, or practicing adequate non-hormonal contraception for at least 3 months prior to and for the duration of study participation. All female subjects will undergo a pregnancy test at screening and at check-in to the clinical study site for every dosing period. The results of the test must be negative for continued participation.
3. Weight must be within 15% of the ideal weight for height and frame, as adopted by the Metropolitan Life Insurance Co., 1993.
4. Qualifying subjects must be in good health and physical condition as determined by a screening medical history obtained within 30 days prior to study start. Subjects should not present with a history of significant past illness expected to affect the investigation.
5. The normal status of subjects will be confirmed by the following procedures:

   1. Laboratory tests (serum chemistry, hematology, urinalysis)
   2. Human immunodeficiency virus (HIV), hepatitis, alcohol, and "drugs of abuse" testing will be done at screening. Results of the HIV, hepatitis, alcohol, and "drugs of abuse" tests must be negative or non-reactive for
   3. Electrocardiogram: A 12-lead electrocardiogram (ECG) will be obtained for all subjects. This ECG must be interpreted by appropriately trained and experienced medical personnel. A subject with an ECG that is not within normal range does not qualify, unless specifically accepted (with comment) by the investigator.
6. Subjects must be able to provide written consent and agree to abide by the study requirements.

Exclusion Criteria:

1. History of alcohol, drug, or narcotic abuse or dependence.
2. Chronic use of tranquilizers, sedatives, aspirin, antibiotics, or other medications.
3. History or presence of major organ dysfunction.
4. History of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorder capable of altering the absorption, metabolism, or elimination of drugs or constituting a risk factor when taking hydromorphone.
5. History of anxiety, tension, severe agitation, psychosis, or mental depression.
6. Family history or diagnosis of epilepsy or other seizure disorder.
7. History of acute abdominal conditions.
8. History of conditions that might contraindicate or require caution be used in the administration of hydromorphone including: renal impairment, hepatobiliary or pancreatic disease, GI obstruction, cardiac disease, obstructive pulmonary disease, acute or severe bronchial asthma, hypercarbia, elevated intracranial pressure, depleted blood volume, paralytic ileus, or allergy to hydromorphone, any opiate agonists, or naltrexone.
9. Administration of any other investigational drug during the 30 days prior to enrollment into the study.
10. Subjects who smoke or have a history of smoking, or use nicotine-containing products.
11. Subjects who have donated blood within 30 days prior to study entry, including that withdrawn during the conduct of any other clinical study.
12. Subjects presenting with acute illness.
13. Subjects who have taken prescription drugs within 14 days or over-the-counter medications (including herbal preparations) within 7 days prior to dosing except for standard daily dose multivitamins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-12; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUCt, AUCinf and Cmax | Two-period crossover with blood samples obtained prior to and following each dose at selected times through 24 hours. Washout period between doses was 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Neuman, MD, Study Director — Mallinckrodt
Locations (1):
- Gateway Medical Research, Saint Charles, Missouri, United States